CLINICAL TRIAL: NCT04280146
Title: Speed Limits: Food Intake and Eating Behaviour of Ultra-processed and Unprocessed Foods
Acronym: Vogue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SEC 2020-11
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Excess Calories
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Subjects are exposed foods for four days. 1 day Ultra processed fast food
  1 day Ultra processed slow foods
  1 day unprocessed fast food
  1 day unprocessed slow food
Who Masked: Participant
Masking Description: Investigate cultural difference on eating behaviour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Degree of food processing (Active Comparator): unprocessed vs ultra-processed foods according to NOVA table.
  Interventions: Behavioral: daily energy intake
- eating rate (Active Comparator): slow vs fast eating rate (kcal/min), manipulated by food form
  Interventions: Behavioral: daily energy intake

INTERVENTIONS:
Behavioral: daily energy intake — Investigate daily energy intake according to eating rate and food processing
  Other Names: eating rate

SUMMARY:
Rationale: Foods that can be eaten at a fast rate - with low mastication effort - lead to shorter orosensory exposure (OSE) per unit of food consumed. This results in a decreased satiation response and higher subsequent food intake. Recent research has shown that participants on a ultra-processed diet have an higher caloric intake and gain body weight compared to those on an unprocessed food diet. In this study the ultra-processed vs. unprocessed meals were classified according to the NOVA classification and matched on caloric content and palatability. The NOVA classification, classifies foods based on the physical, biological and chemical processes that occur after foods are separated from nature, and before they are consumed or used in the preparation of dishes and meals.

However, it remains unclear whether the found increase in food intake of ultra-processed foods is due to industrial processing or because of a difference in eating rate at which the (ultra-)processed foods can be consumed.

Objective: The objective of this study is to determine the independent and additive effects of industrial food processing (according to the NOVA classification) and eating rate on satiation.

Study design: The study has a 2x2 randomized crossover design. All participants receive 4 treatments and are their own control.

Study population: Healthy adults (n=60) between 18-55 years old with a BMI between 18.5-27 kg/m2.

Intervention: Participants will join 4 test days during which they receive 3 main test meals (breakfast, lunch, dinner) and in-between meals snacks according to one of the 4 diets. The 4 diets of this study are: 1) unprocessed, slow eating rate 2) unprocessed, fast eating rate 3) ultra-processed, slow eating rate 4) ultra- processed, fast eating rate. During eating and before and after eating the weight of the plate will be measured to determine intake. Additionally, participants will be recorded on video to determine eating behaviour (number of bites, chews and oral processing duration). The order in which participants will receive the diets will be randomized. The evening before and during each test day participants will keep a food and exercise diary.

Main study parameters/endpoints: The main study outcomes are food intake during the three main meals and during snack time. Secondary outcomes are, eating behaviour characteristics measured by video (eating rate (g/min and bites/min), number of chews (chews/bite and chews/gram), bite size (gram/bite), oral processing duration (seconds), appetite (hunger, fullness, desire to eat, desire to eat sweet, desire to eat savoury, prospective consumption) and sensory characteristics (liking (taste + smell), desire to eat the meal, expected satiation, sweet, savoury, smoothness, chewiness, thickness) of the meals.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk associated with participation is small and the burden can be considered as moderate. The knowledge obtained may be used to develop products or strategies that enhance healthy choices and eating behaviour and consequently help prevent overweight and obesity. We consider the knowledge obtained and possible implications of this study to outweigh the individual burden.

DETAILED DESCRIPTION:
1. OBJECTIVE

   The objective of this study is to determine the independent and additive effects of industrial food processing (according to the NOVA classification) and eating rate on satiation

   Hypothesis:

   We expect that a slow eating rate decreases food intake per main meal and over the course of the day, independent of industrial processing.
2. STUDY DESIGN

The study has a 2x2 randomized crossover design; all participants receive each treatment and are their own control (within subject effects). See table 1 for an overview of a test day.

The 4 conditions of this study are:

1. unprocessed slow eating rate
2. unprocessed fast eating rate
3. ultra- processed slow eating rate
4. ultra- processed fast eating rate

   Timing Activity/Instruction Throughout study period • No use of drugs. Medication use + illness should be reported Previous day • Keep a food and exercise diary
   * No intensive exercise (only regular speed walking and biking)
   * No alcoholic drinks Evening Preceding test day • Same evening meal of own choice between 18.00-19.30
   * Not allowed to eat or drink (any caloric) after 10 p.m. except for water Morning of test day • Not allowed to eat or drink anything besides a glass of water
   * Keep food and exercise diary Breakfast • Check adherence to study rules
   * Check food diary
   * Give instructions test day
   * Seated at table
   * Appetite questionnaire
   * Sensory questionnaire
   * Eat meal [one of 4 conditions- randomized] *Record intake

     *Record eating behaviour
   * Reason to end the meal + Appetite questionnaire
   * Sensory questionnaire Break • Give instructions snacks [no need to eat all, as much or as little as you want, not allowed to eat anything else, allowed to drink water thee and coffee without milk or sugar. Participants will be asked to bring back leftovers.

   Lunch • Check adherence to study rules
   * Check food diary
   * Give instructions
   * Seated at table
   * Appetite questionnaire
   * Sensory questionnaire
   * Eat meal [one of 4 conditions- randomized] *Record intake

     *Record eating behaviour
   * Reason to end the meal + Appetite questionnaire
   * Sensory questionnaire Break • Give instructions snacks [no need to eat all, as much or as little as you want, not allowed to eat anything else, allowed to drink water thee and coffee without milk or sugar. Participants will be asked to bring back leftovers.

   Dinner • Check adherence to study rules • Check food diary • Give instructions • Seated at table • Appetite questionnaire

   • Sensory questionnaire

   • Eat meal [one of 4 conditions- randomized]

   *Record intake
   * Record eating behaviour

     * Reason to end the meal + Appetite questionnaire
     * Sensory questionnaire Break • Give instructions snacks [no need to eat all, as much or as little as you want, not allowed to eat anything else, allowed to drink water thee and coffee without milk or sugar. Participants will be asked to bring back leftovers.

   Table 1. Study (pre-) day overview. Participants join four test days during which they eat ad libitum of 3 main test meals (breakfast, lunch, dinner) in between meals they receive snacks.

3. STUDY POPULATION

3.1 Population (base)

Participants will be recruited from Wageningen and surroundings. Healthy (self-report), normal to slightly overweight (18.5-30 kg/m2) men and women between 18-55 years old will be included. Participants have to be able to understand and speak English (self-report), because of the sensory questionnaire and appetite questionnaire which will be in English and have difficult direct translations to Dutch. As 90% of the people that show interest in the study are university students this should not be a problem (i.e. limiting the number of people that can be included in the study). The BMI range is based on the average BMI in the Netherlands, which is 25 kg/m2 but around 50% of the Dutch population is overweight. To be able to include sufficient subjects we therefore choose to widen the BMI range and include people up to a BMI of 30 kg/m2 (20). Due to the within subject design this will not influence the outcome of the study, but results will be more generalizable to people with an average weight.

3.2 Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following inclusion criteria:

* Between 18-55 years old at the day of inclusion
* Able to understand and speak English fluently or without difficulty (self-report)
* BMI 18.5-30 kg/m2 - measured by the researchers at the end of information meeting (after signing informed consent)
* Good general health and appetite (F1 questionnaire self-report)
* Commonly (5 out of 7 week days) eating three meals a day every day around approximately the same times. (This is a Self-report question; see F1 questionnaire).

3.3 Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Difficulties with swallowing, chewing and or eating in general
* Suffering from an endocrine or eating disorder, gastrointestinal illness or illness of the thyroid gland, respiratory disease or diabetes.
* Having taste or smell disorders (self-report)
* Braces (not including a dental wire) or oral piercing
* Smoking
* Consuming on average more than 21 glasses of alcohol per week (21)
* Not willing to stop using drugs during the study period (from inclusion till last test session)
* Use of medication that may influence study outcomes (self-report)
* Allergies or intolerance to any ingredient of the test meals or snacks
* Not willing to eat the test food because of eating habits or believes.
* Following a vegetarian or vegan diet
* Lactose intolerant
* Men having facial hair such as a beard as facial movements cannot be analysed.
* Followed an energy restricted diet during the last 2 months
* Gained or lost 5 kg of body weight over the last half year
* High restrained eater according to the Dutch Eating Behaviour Questionnaire (men: score>2.9)*. * This exclusion criterion will not explicitly be communicated to the participants to prevent desirable answers.
* Signed up for participating in another research study
* Employee of Human Nutrition department of Wageningen university
* Thesis student or intern at the chair group of Sensory Science and Eating Behaviour Human Nutrition (WUR).
* Intensive exercising more than 8 hours per week
* Low score (< -1) for liking the test foods on a nine point likert scale based on pictures of the food items.
* Unfamiliar with the test foods (self report).

3.4 Screening during Information meeting

People interested in participating in the study can send an email to the investigator indicating that they would like to join the study. After that, participants will receive an invitation for the information meeting and a pdf of the information brochure by email. During the information meeting prospective participants receive information about the procedure, design and measurements of the study through an oral presentation. Participants will not be informed about the study's purpose. Participants will be told that we are interested in eating behaviour differences between cultures. It will not be explained specifically that the main interest is the amount eaten during the ad libitum test meals as this may influence the results. Participants will be informed about the specific parameters of interest when the study is finished by email. After receiving the information participants are free to sign their informed consent.

After signing informed consent, participants will be asked to fill in the Dutch Eating Behaviour Questionnaire (DEBQ: 33 questions) together with other in-exclusion criteria (health) questions.

After filling in the questionnaires, participants will be asked to rate liking and familiarity of the test food meals based on pictures and taste and rate liking of the snacks on a nine point hedonic and visual analogue scale (VAS). Based on the in- and exclusion criteria participants are invited for the test days.

4. Sample size

The main outcome of interest is satiation measured through ad libitum intake of test meals.

Based on our previous studies that had the same outcome we need to include 60 participants to be able to find a 10% difference between study treatments.

5. Study measures and meals

5.1 measurements study

During test meals (breakfast, lunch, dinner) participants eat ad libitum of a test meal according to one of the four conditions ; unprocessed slow eating rate, unprocessed fast eating rate, ultra-processed slow eating rate, ultra-processed fast eating rate. During the meal intake will be measured using a weighing scale hidden in a tray and video recordings will be made to determine eating behavior. Before and after the test meals participants will be asked to rate sensory and appetite questions.

General Health and well-being questionnaire The general health and well-being questionnaire of the human nutrition department will be used to ask subjects about their health and well-being (since their last session) at the start of the test day.

Appetite, sensory and well-being variables

Participant will answer an appetite questionnaire. They will rate hunger, fullness, thirst, desire to eat, desire to eat sweet/savoury, and general prospective consumption on a 100-mm visual analogue scale (VAS) ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line.

Appetite Factors:

Hunger Fullness Desire to eat Desire to eat sweet Desire to eat savoury Prospective consumption

In addition, participants will rate first the sensory/hedonic attributes of the meal on a 100-mm VAS scale ranging from 'not at all' to 'extremely' with anchors at the beginning and end of the line.

Sensory/hedonic characteristics:

Asked only before the meal:

Expected satiation Desire to eat the meal (visually)

Asked before and after the meal:

Liking smell Liking taste/flavour Desire to eat the meal (based on tasting)

Besides these questions we will also let participants indicate their reason to stop eating, If their reason is not indicated they have to choose the most appropriate one:

* I was full
* I got bored with the texture
* I got bored with the flavour
* I got tired chewing
* I ate the portion I would normally eat

In addition we will ask participants to rate wellbeing parameters.

* Nausea
* General wellbeing

Video recordings

During the ad libitum eating meals participants will be video recorded. A digital camera will be positioned in front of the subject (face-on) where the lower frame will be in line with the shoulders, the upper frame wil be above the top of the cranium and the sides at shoulder width. Participants will be instructed to look straight into the webcam and not to make excessive head movements. Data will be analysed manually with use of Observer Noldus. Recordings will be analysed in a random order. Beforehand defined indicators are: number of bites, total eating duration, eating duration per bite, number of masticatory cycles per bite. Application of this technique to chewing of gel-like model foods has shown that it is possible to separate subjects based on their chewing behaviour (28-31). Permission to record the participant and save and use the video for this study's purpose will be asked on the informed consent form.

5.1 NOVA classification of unprocessed, processed (culinary), processed and ultra-processed foods.

Group 1 Unprocessed Group 2 Processed (culinary) Group 3 Processed Group 4 Ultra-processed Fruit Oils Canned vegetables Soft drinks Leaves Butter Bottled vegetables Packed snacks Stems Lard Canned legumes Candies/ chocolate Seeds Sugar Bottled legumes Mass produced breads Roots Salt Fruit in syrup Cookies Meat Tinned fish in oil Pastries Eggs Bacon Cakes Milk Ham Margarine Fungi Pastrami Sweetened breakfast cereals Algea Smoked fish Fruit yoghurt water Simple cheeses Energy drinks Freshly baked bread Pre-prepared meat Cheese Pasta/noodles Pizza Nugget Burgers Hot dogs Sausages Instant soups Dessert

6. Withdrawal of individual subjects Subjects may discontinue the trial at any moment without the obligation to state the reason for discontinuation. Subjects may be withdrawn from the study by the principal investigator if they do not comply with the rules and regulations of the study. Subjects may be withdrawn from the study by the medical supervisor in case of reported serious adverse events or in case of other medical/social/psychological events as evaluated by the medical investigator and discussed with the principal investigator.

6.1 Replacement of individual subjects after withdrawal A total of 60 participants will be included and we will aim to have 5 participants on the reserve list to participate if participants drop-out during the first week of the study.

7. Incentives Participants do not receive reimbursement for the information meeting as we expect not to be able to include many of the participants due to the extensive in- and exclusion criteria. For completing the entire study (four test sessions) participants receive €100, - euro. Participants receive €20, - reimbursement per session if they drop out of the study and participants receive an additional €20, - when completing the entire study. The reimbursement is calculated (+/- 10%) based on guidelines of the Human Nutrition department of Wageningen University.

8. Handling and storage of data and documents

All the gathered data will be handled confidential through coding, except for the video's where the participant will be recognizable. All subjects will receive a unique code, and only the project leader and investigators will have the key. Confidentially will be clearly communicated to all participants .The personal data will be stored in a digital database on an intern network which is protected by a personal password. The password is only known by the investigators. The key to the personal information will be kept until 5 years after the results of the study are published and is only known by the project leader and coordinating researcher. All other data will be kept for 15 years after the results of the studie are published. No names of the participants will be used in the publication of this study.

The video recordings will be stored on the W: drive of the department, only the researchers directly involved in the study are given access to this drive when login on their account including password. Videos will be labelled with a unique code, not traceable to the participant, however to obtain mastication parameters it is necessary to have recordings of the entire head of the participant; therefore video's will not be anonymous. The videos will be analysed by the project leader, principle investigator and possible research assistant and or BSc/MSc thesis/internship students but will be handled confidentially. All researchers and assistant involved in the study will sign a confidentiality form. The videos will be kept for 5 years after the results of the study are published. Permission of the subjects will be asked to be able to do so, at the informed consent form. Videos will solely be used for the analysis as described in this protocol. Videos will not be used for presentation purposes only in case the participant gives verbally and in written permission to do so.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-55 years old at the day of inclusion

  * Able to understand and speak English fluently or without difficulty (self-report)
  * BMI 18.5-30 kg/m2 - measured by the researchers at the end of information meeting (after signing informed consent)
  * Good general health and appetite (F1 questionnaire self-report)
  * Commonly (5 out of 7 week days) eating three meals a day every day around approximately the same times. (This is a Self-report question; see F1 questionnaire).

Exclusion Criteria:

* Difficulties with swallowing, chewing and or eating in general
* Suffering from an endocrine or eating disorder, gastrointestinal illness or illness of the thyroid gland, respiratory disease or diabetes.
* Having taste or smell disorders (self-report)
* Braces (not including a dental wire) or oral piercing
* Smoking
* Consuming on average more than 21 glasses of alcohol per week (21)
* Not willing to stop using drugs during the study period (from inclusion till last test session)
* Use of medication that may influence study outcomes (self-report)
* Allergies or intolerance to any ingredient of the test meals or snacks
* Not willing to eat the test food because of eating habits or believes.
* Following a vegetarian or vegan diet
* Lactose intolerant
* Men having facial hair such as a beard as facial movements cannot be analysed.
* Followed an energy restricted diet during the last 2 months
* Gained or lost 5 kg of body weight over the last half year
* High restrained eater according to the Dutch Eating Behaviour Questionnaire (men: score>2.9)*. * This exclusion criterion will not explicitly be communicated to the participants to prevent desirable answers.
* Signed up for participating in another research study
* Employee of Human Nutrition department of Wageningen university
* Thesis student or intern at the chair group of Sensory Science and Eating Behaviour Human Nutrition (WUR).
* Intensive exercising more than 8 hours per week
* Low score (< -1) for liking the test foods on a nine point likert scale based on pictures of the food items.
* Unfamiliar with the test foods (self report).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Energy intake | 1 day
  Daily energy intake

CONTACTS AND LOCATIONS:
Overall Officials: Dieuwerke P Bolhuis, PhD, Principal Investigator — Wageninge University
Locations (1):
- Wageningen University, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lasschuijt M, Camps G, Mars M, Siebelink E, de Graaf K, Bolhuis D. Speed limits: the effects of industrial food processing and food texture on daily energy intake and eating behaviour in healthy adults. Eur J Nutr. 2023 Oct;62(7):2949-2962. doi: 10.1007/s00394-023-03202-z. Epub 2023 Jul 14. PMID 37452167